CLINICAL TRIAL: NCT06392386
Title: An Open-label, Uncontrolled Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Safety, and Activity of Efgartigimod PH20 SC in Participants From 2 to Less Than 18 Years of Age With Generalized Myasthenia Gravis
Brief Title: A Study of Efgartigimod PH20 SC in Children Between 2 and Less Than 18 Years of Age With Generalized Myasthenia Gravis
Acronym: ADAPT Jr SC
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARGX-113-2207; 2023-506159-12-00 (EU CTIS Number)
Record Dates: First submitted 2024-04-26; First posted 2024-04-30 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Generalized Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Efgartigimod PH20 SC (Experimental): Participants aged 12 to <18 years receiving efgartigimod PH20 SC treatment
  Interventions: Biological: Efgartigimod PH20 SC

INTERVENTIONS:
Biological: Efgartigimod PH20 SC — Subcutaneous injections

SUMMARY:
The purpose of this study is to measure the pharmacokinetics (PK), pharmacodynamics (PD), safety, tolerability, and immunogenicity of efgartigimod PH20 SC in pediatric participants with gMG aged 2 to <18 years. The primary goal is to confirm an appropriate dose of efgartigimod PH20 SC for pediatric patients using PK and PD results from this study. Participants will receive injections of efgartigimod PH20 SC and will be monitored for safety until the end of the study. At the end of the follow-up period, eligible participants may roll over to an open-label extension (OLE) study.

The participants will be in the study for up to 14 weeks.

ELIGIBILITY:
Inclusion Criteria:

* The participant (and/or their legally authorized representative) understands the requirements of the study and is capable of providing written informed consent/assent and complying with protocol requirements
* The participant is aged 2 to <18 years at the time of informed consent/assent
* The participant has been diagnosed with generalised Myasthenia Gravis that is supported by a physical examination and confirmed seropositivity for anti-acetylcholine receptor antibodies
* The participant has had an unsatisfactory response to immunosuppressants, corticosteroids, or acetylcholinesterase inhibitors but is on stable concomitant MG therapy. If receiving corticosteroids and/or immunosuppressants, must be on a stable dose for ≥1 month before screening
* The participant agrees to use birth control consistent with local regulations and people of child-bearing potential must have a negative blood pregnancy test at screening and a negative urine pregnancy test before receiving the study drug

Exclusion Criteria:

* Is a female adolescent of child-bearing potential who is pregnant and/or lactating or intends to become pregnant during their participation in the study
* Has worsening muscle weakness secondary to a concurrent infection or as a result of a medication
* Has a documented lack of clinical response to plasma exchange (PLEX)
* Received a live or live-attenuated vaccine within <4 weeks before screening
* Received a thymectomy within 3 months before screening or is planning to get a thymectomy during their participation in the study
* Has a known autoimmune disease or any medical condition that would interfere with an accurate assessment of clinical symptoms of generalised Myasthenia Gravis or puts the participant at undue risk
* History of malignancy, cancer, unless considered cured by adequate treatment with no evidence of recurrence for ≥3 years. Adequately treated participants with the following cancers can be included at any time: Basal cell or squamous cell skin cancer, Carcinoma in situ of the cervix, Carcinoma in situ of the breast, Incidental histological findings of prostate cancer
* Clinically significant active infection that is not sufficiently resolved in the investigator's opinion or positive serum test at screening for active infection with any of the following: Hepatitis B virus (HBV), Hepatitis C virus (HCV), HIV
* Has a positive PCR test for SARS-CoV-2 at screening
* Has/had a clinically significant disease, had recent major surgery (within 3 months of screening) or intends to have major surgery during the study, or has/had any other medical condition that, in the investigator's opinion, would confound the results of the study or put the participant at undue risk
* Has received a different study drug in another clinical study within <12 before screening
* Is currently participating in another interventional clinical study
* Has previously participated in an efgartigimod clinical study and received at least one dose of study drug
* Has a known hypersensitivity to study drug or any of its excipients
* Has a history of or current episode of alcohol, drug, or medication abuse as assessed by the investigator
* Use of some medications before screening (more information is found in the protocol)

The complete list of exclusion criteria can be found in the protocol.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2024-06-28 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Efgartigimod serum concentrations as input for compartmental, model-driven analysis to determine age and size dependency of Clearance (CL) | Up to 12 weeks
Efgartigimod serum concentrations as input for compartmental, model-driven analysis to determine age and size dependency of Volume Distribution (Vd) | Up to 12 weeks
Total G immunoglobulins (IgG) levels as input for pharmacokinetics (PK)/pharmacodynamics (PD) modelling analysis | Up to 12 weeks
Anti-acetylcholine receptors antibodies (AChR-Ab) as input for pharmacokinetics (PK)/ pharmacodynamics (PD) modelling analysis | Up to 12 weeks

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 14 weeks
Severity of adverse events (AEs) | Up to 14 weeks
Incidence of serious adverse events (SAEs) | Up to 14 weeks
Severity of serious adverse events (SAEs) | Up to 14 weeks
Incidence of adverse events of special interest (AESI) | Up to 14 weeks
Severity of adverse events of special interest (AESI) | Up to 14 weeks
Efgartigimod serum concentrations | Up to 12 weeks
Absolute values of total Immunoglobulin G (IgG) from blood samples | Up to 12 weeks
Change from baseline values of total Immunoglobulin G (IgG) from blood samples | Up to 12 weeks
Percentage change from baseline values of total Immunoglobulin G (IgG) from blood samples | Up to 12 weeks
Absolute values of anti-acetylcholine receptor antibodies (AChR-Ab) from blood samples | Up to 12 weeks
Change from baseline values of anti-acetylcholine receptor antibodies (AChR-Ab) from blood samples | Up to 12 weeks
Percentage change from baseline values of anti-acetylcholine receptor antibodies (AChR-Ab) from blood samples | Up to 12 weeks
Incidence of anti-drug antibodies (ADAs) against efgartigimod in serum samples | Up to 12 weeks
Prevalence of anti-drug antibodies (ADAs) against efgartigimod in serum samples | Up to 12 weeks
Incidence of antibodies against rHuPH20 in serum samples | Up to 12 weeks
Prevalence of antibodies against rHuPH20 in serum samples | Up to 12 weeks
Absolute value of total Myasthenia Gravis Activity of Daily Living (MG-ADL) score, appropriate for pediatric use | Up to 12 weeks
  Minimum value: 0 (no impairment); Maximum value: 24 (highest impairment)
Change from baseline of total Myasthenia Gravis Activity of Daily Living (MG-ADL) score, appropriate for pediatric use | Up to 12 weeks
  Minimum value: 0 (no impairment); Maximum value: 24 (highest impairment)
Absolute value of Quantitative Myasthenia Gravis (QMG) score | Up to 12 weeks
  Minimum value: 0 (no impairment); Maximum value: 39 (most severe impairment)
Change from baseline of Quantitative Myasthenia Gravis (QMG) score | Up to 12 weeks
  Minimum value: 0 (no impairment); Maximum value: 39 (most severe impairment)
Absolute value of EuroQoL 5 Dimensions Youth (EQ-5D-Y) score | Up to 12 weeks
Change from baseline value of Neuro-QoL Pediatric Fatigue Score | Up to 12 weeks
Change from baseline value of EuroQoL 5 Dimensions Youth (EQ-5D-Y) score | Up to 12 weeks
Change from baseline value of Clinical Global Impression of Improvement (CGI-I) | Up to 12 weeks
Changes in protective antibody titers to vaccines | Up to 12 weeks

CONTACTS AND LOCATIONS:
Locations (20):
- United States (3):
  - Carolinas HealthCare System Neurosciences Institute - Neurology, Charlotte, North Carolina
  - Neurology Rare Disease Center, Denton, Texas
  - University of Virginia, Charlottesville, Virginia
- UZ Gent, Ghent, Belgium
- Childrens Hospital of Eastern Ontario, Ottawa, Canada
- Czechia (2):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Ostrava, Ostrava
- AP-HM- Hôpital de La Timone, Marseille, France
- Universitätsklinikum Essen, Essen, Germany
- Israel (3):
  - Hadassah Medical Center- Ein Kerem, Jerusalem
  - Schneider Children's Medical Center of Israel, Petah Tikvah
  - Tel Aviv Sourasky Medical Center Ichilov, Tel Aviv
- Istituto G Gaslini Ospedale Pediatrico IRCCS, Genova, Italy
- Leiden University Medical Center, Leiden, Netherlands
- Poland (3):
  - Uniwersyteckie Centrum Kliniczne w Gdansku, Gdansk
  - Neurologia Śląska Centrum Medyczne, Katowice
  - Centralny Szpital Kliniczny - Uniwersyteckie Centrum Kliniczne WUM, Warsaw
- Hospital Universitari i Politecnic La Fe de Valencia, Valencia, Spain
- Hôpital Nestlé, Lausanne, Switzerland
- Oxford Children's Hospital, Oxford, United Kingdom